CLINICAL TRIAL: NCT06275685
Title: Forecasting Seizures Using IntelliGent Wearable Technology for Health Tracking
Acronym: Foresight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Empatica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIP-0001510
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Epilepsy; Seizure
Keywords: forecasting
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): The control arm will receive multi-day visualizations of their sensor derived data but not receive SeizureWise
  Interventions: Device: Multi-day Visualizations
- Personalized seizure risk score (Experimental): The personalized seizure risk score arm will receive multi-day visualization of their sensor derived data and also SeizureWise, an investigational algorithm which enables forecasting of future seizure probabilities based on the pattern and frequency of previous generalized tonic-clonic seizure (GTCS) events, as well as changes in physiological and behavioral variables
  Interventions: Device: SeizureWise algorithm; Device: Multi-day Visualizations

INTERVENTIONS:
Device: SeizureWise algorithm — An investigational algorithm which enables forecasting of future seizure probabilities based on the pattern and frequency of previous generalized tonic-clonic seizure (GTCS) events, as well as changes in physiological and behavioral variables
  Arms: Personalized seizure risk score
Device: Multi-day Visualizations — Multi-day visualizations of sensor derived data

SUMMARY:
The goal of this interventional study is to develop a personalized seizure risk forecast tool in people with epilepsy.

The main questions it aims to answer are:

* can we develop a future seizure probabilities tool that is more accurate than chance based on the pattern and frequency of previous generalized tonic-clonic seizure (GTCS) events, as well as changes in physiological and behavioral variables.
* does this tool improve the lives of people with epilepsy?

Researchers will compare a group that does not have access to the forecast tool to a group that does and see if it is accurate and if people with it report that it improved their quality of life.

DETAILED DESCRIPTION:
The primary goal of the study is to demonstrate the accuracy of SeizureWise in predicting the timing of future convulsive seizures using data collected by the wearable EmbracePlus device and data provided by patients with GTCS monitored in outpatient settings.

The secondary goals are:

to assess the clinical impact of SeizureWise on quality of life (QoL), psychological health indicators, and economic and clinical outcomes to assess the clinical impact of visualizing behavioral and physiologic data without forecasting predictions on quality of life (QoL), psychological health indicators, and economic and clinical outcomes

A non-significant risk, open-label, prospective, randomized clinical investigation designed to evaluate the ability of SeizureWise to forecast GTCS occurrence and to assess impact on QoL and seizure management outcomes.

The study will include two phases during which an algorithm based on sensor derived physiological measures is developed and tested with output blinded to the participant. In a final phase participants will be randomized to two arms, one of which will have access to a seizure forecasting risk score.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be diagnosed with or be at risk of epilepsy
* Subjects or their parents or guardians must understand and consent to be in the study;
* Subjects or their parents or guardians must be able to read and communicate in English;
* Subjects or their parents or guardians must be willing and able to comply with study procedures and duration;
* Subjects must have a wrist circumference suitable for wearing the EmbracePlus device.

Exclusion Criteria:

* Subjects, or their parents or guardians for minor study participants, who do not understand the study and the risks;
* Subjects, or their parents or guardians for minor study participants, who are either physically or cognitively incapable of performing study activities (e.g. filling in surveys and daily e-diary);
* Subjects who would be placed at undue medical risk associated with any procedure called for in the protocol; or
* Subjects that are Empatica employees and actively participated in the development of this protocol or development of the Seizure Wise algorithms.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of SeizureWise | 2 years
  Percentage of patients with (1) sensitivity of high-likelihood warnings greater than 60% and (2) superior to a rate-matched forecast (or superior baselining method) at the end of Phase 2.

SECONDARY OUTCOMES:
Change in QoL and psychological health indicators using the Quality of life in epilepsy (QOLIE-10-P) | 2 years
  Changes in QoL and psychological health indicators pre- and post-Phase 3 (cross-arm and intra-arm comparisons. This will be assessed using the QOLIE-10-P and scored according to these guidelines https://www.aan.com/siteassets/home-page/policy-and-guidelines/quality/quality-measures/epilepsy-and-seizures/qolie10p-scoring.pdf
Qualitative assessment of multi-day visualizations | 2 years
  Patient-reported qualitative assessment of multi-day visualizations to the patient during Phase 3 (both arms). This will be assessed using a custom survey and a qualitative analysis of the scores will be performed between start of phase 3 (with no visualizations) and during and at the end of phase 3 when visualizations have been provided to the user.
Stress level with visualizations using the brief epilepsy anxiety survey instrument (brEASI-8) | 2 years
  Quantitative patient report of stress level pre- and post- forecast visualization during Phase 3 in the intervention arm. This will be assessed using brEASI-8 where a lower score indicates a lower stress level.
Modifiable behavior change | 2 years
  Adjustment in modifiable behaviors during Phase 3 based on multi-day visualizations (boths arms) and forecast outputs (intervention arm). This will be assessed using a custom survey and a qualitative analysis will be performed that looks at participants behaviors before and after receiving visualizations and SeizureWise.
Accuracy of SeizureWise low-likelihood forecast | 2 years
  Percentage of time in a low-likelihood forecast category during which no seizure event occurs during Phase 2.
Accuracy of SeizureWise high-likelihood forecast | 2 years
  Percentage of time in a high-likelihood forecast category during which a seizure event occurs during Phase 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Empatica, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No